CLINICAL TRIAL: NCT04610450
Title: The Performance of a Robot-assisted Minimally Invasive Direct Cochlear Access for Cochlear Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCI-NEXT
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-05

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RCI-BE-10 (Experimental): Robot assisted cochlear implant surgery.
  Interventions: Device: HEARO; Device: OTOPLAN

INTERVENTIONS:
Device: HEARO — Robotic system for otological procedures
Device: OTOPLAN — Otological surgical planning software

SUMMARY:
The cochlear implant is a neural prosthesis and has been the gold standard treatment for severe to profound sensorineural hearing loss over several decades. The surgical procedure for cochlear implantation aims to atraumatically insert the electrode array of the cochlear implant into the cochlea. However, due to the location of the cochlea inside the skull, the surgeon is required to create an access from the surface of the temporal bone to the cochlea (inner ear). In conventional methods, this access is acquired by removal of portions of the mastoid bone through a mastoidectomy and posterior tympanotomy. The outcome and success of the conventional procedure varies due to mainly two factors: surgeon skill and subject anatomical variation. To overcome these variables toward a more consistent and less invasive cochlear implantation surgery, the development of robotic and image guided cochlear implantation has taken place. This study primarily aims to explore the performance of robotic cochlear implantation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for CI surgery according to clinical routine
* Subjects who will receive a cochlear implant
* Signed and dated informed consent form

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Age under 18 years
* Pregnancy
* Distance of the planned trajectory to the facial nerve is < 0.4 mm as per screening CT scan
* Distance of the planned trajectory to the chorda tympani is < 0.3 mm as per screening CT scan
* A safe inner ear access cannot be planned for preservation of RW membrane and cochlear structures
* Individuals where image guidance or robotic procedures are not indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Relative ratio of successful electrode array insertions through the drilled direct cochlear access with the HEARO procedure to the total HEARO procedures. | day 0
  The primary outcome measure of this study is to explore the relative ratio of the successful electrode array insertions into the cochlea through the drilled direct cochlear access with the HEARO procedure to the total HEARO procedures. Aborted or converted procedures count as procedure in which insertion through the direct cochlea access was not possible. The results will be expressed in relative numbers and in percentage.

SECONDARY OUTCOMES:
Electrode array insertion outcome | day 0
  The angular insertion depth (in degrees) will be evaluated.
Electrode array insertion outcome | day 0
  The number of inserted electrode contacts will be evaluated.
Electrode array insertion outcome | day 0
  The surgical outcome (categories: nominal, tip-fold over or scalar deviation) will be evaluated.
Insertion depth prediction accuracy | day 0
  The insertion depth prediction accuracy as the difference between the estimated insertion depth of the electrode at the planning and the actual insertion depth.
Absolute angular accuracy of the drilled tunnel access | day 0
  The absolute in-plane and out-plane accuracy of the drilled tunnel is measured as the angular deviation between the planned trajectory in-plane and out-plane angles and the actual drilled angles from the intra-op image.
Absolute lateral accuracy of the drilled tunnel at the facial recess | day 0
  The absolute lateral accuracy of the drilled tunnel to the facial nerve and chorda tympani is measured as the difference between the planned trajectory and the actual drilled trajectory distance.
Absolute lateral accuracy of the drilled tunnel at the target | day 0
  The absolute lateral accuracy of the drilled tunnel is measured as the distance between the planned target trajectory position and actual target of the drilled trajectory position.
Ratio of the round window membrane preservation during the inner ear access | day 0
  The ratio of the visibility of round window membrane surface at the robotic inner ear access by visual inspection. This will be assessed as subjective evaluation by the surgeon.
Timing of the HEARO procedure | day 0
  The timing of the different steps of the HEARO procedure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Caversaccio, Prof. Dr., Principal Investigator — University Hospital Bern (Inselspital)
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No